CLINICAL TRIAL: NCT06090916
Title: Malnutrition Screening and Nutrition Optimization to Improve Outcomes in Patients With Unresectable Pancreatic Cancer
Brief Title: Malnutrition Screening and Dietary Intervention to Improve Nutrition Outcomes in Patients With Unresectable Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Silicon Valley Community Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-000208; NCI-2023-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Stage III Pancreatic Cancer; Pancreatic Adenocarcinoma Non-resectable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Diet Therapy; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM I (Standard of care) (Active Comparator): Patients receive standard nutrition care and record dietary intake and physical activity using Myfitness Pal smartphone application on study.
  Interventions: Other: Best Practice; Other: Medical Chart Review; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration
- ARM II (Dietary intervention) (Experimental): Patients undergo malnutrition screening with a registered dietician at baseline and participate in 12 weekly nutrition support sessions and those at moderate to high risk for malnutrition receive a personalized diet prescription on study. Patients also record dietary intake and physical activity using Myfitness Pal smartphone application on study.
  Interventions: Other: Dietary Intervention; Other: Medical Chart Review; Other: Medical Device Usage and Evaluation; Other: Nutritional Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard nutrition care
  Other Names: standard of care; standard therapy
  Arms: ARM I (Standard of care)
Other: Dietary Intervention — Participate in weekly support sessions with diet prescription
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: ARM II (Dietary intervention)
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Medical Device Usage and Evaluation — Record dietary and physical activity using MyFitnessPal smartphone app
Other: Nutritional Assessment — Undergo malnutrition screening
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
  Arms: ARM II (Dietary intervention)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares the effect of malnutrition screening and dietary intervention to standard nutrition care on patients with pancreatic cancer that cannot be removed by surgery (unresectable). Fewer than 20% of patients diagnosed with unresectable pancreatic cancer do not survive one year after diagnosis so treatment often focuses on improving quality of life. Many patients experience increasing pain, nausea, vomiting, loss of appetite, weight loss and weakness. Behavioral interventions use techniques to help patients change the way they react to environmental triggers that may cause a negative reaction. Screening for inadequate nutrition (malnutrition) and providing weekly nutritional support may be effective methods to improve nutritional status and improve overall quality of life for patients with unresectable pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the quality of life of subjects after 12 weeks between the intervention group with nutrition optimization with dietary prescription and nutrition support in comparison to standard care.

II. To compare the frequency of hospitalization and length of stay (LOS) after 12 weeks between the intervention group with nutrition optimization with dietary prescription and nutrition support in comparison to standard care.

III. To compare the subject's functional status, body weight and dietary intake after 12 weeks between the intervention group with nutrition optimization with dietary prescription and nutrition support in comparison to standard care.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard nutrition care and record dietary intake and physical activity using Myfitness Pal smartphone application on study.

ARM II: Patients undergo malnutrition screening with a registered dietician at baseline and participate in 12 weekly nutrition support sessions and those at moderate to high risk for malnutrition receive a personalized diet prescription on study. Patients also record dietary intake and physical activity using Myfitness Pal smartphone application on study.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable pancreatic adenocarcinoma, receiving either 1) no chemotherapy, 2) 1st cycle of chemotherapy, or 3) greater than 1 cycle of chemotherapy if the patient's prognosis is greater than 6 months as determined by oncology collaborators
* Life expectancy of greater than 3 months and a Karnofsky performance score of 60 or more
* Adults >= 18 years old male or female

Exclusion Criteria:

* Ascites requiring paracentesis for symptom improvement
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values greater than 5 times the upper limit of normal
* Creatinine value greater than 2.0 for men and 1.5 for women
* Uncontrolled pain
* Uncontrolled nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured comparing changes in outcomes between study arms | After 12 weeks
  Measured using short form 36. A two-sample t-test comparing changes from baseline in each of the outcomes between study arms used to estimate power
Frequency of hospitalizations | After 12 weeks
  Hospitalization defined as any stay in the hospital > 24 hours. A two-sample t-test comparing changes from baseline in each of the outcomes between study arms used to estimate power
Length of hospital stay | After 12 weeks
  Length of stay determined by the number of days of hospitalization including the date of admission and not including the day of discharge from the hospital. A two-sample t-test comparing changes from baseline in each of the outcomes between study arms used to estimate power
Functional status using Karnofsky performance score | After 12 weeks
  The Karnofsky Performance Status (KPS) is a standardized measure used to assess a patient's ability to perform everyday tasks. It ranges from 0 to 100, with higher scores indicating better function.
Percent change in body weight | Baseline to after 12 weeks
  Collected from patient medical record. A two-sample t-test comparing changes from baseline in each of the outcomes between study arms used to estimate power
Average daily steps | After 12 weeks
  Daily steps recorded using MyfitnessPal. A two-sample t-test comparing changes from baseline in each of the outcomes between study arms used to estimate power
Calorie intake from Myfitness Pal | After 12 weeks
  Food intake collected every 4 weeks and uploaded into patients medical record via patient portal. A two-sample t-test comparing changes from baseline in each of the outcomes between study arms used to estimate power

CONTACTS AND LOCATIONS:
Overall Officials: ZhaoPing Li, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States